CLINICAL TRIAL: NCT05386420
Title: A Single-center, Randomized, Parallel Controlled, Double-blind Clinical Trial Designed to Evaluate the Efficacy and Safety of Hymecromone Tablets in Subjects Diagnosed With COVID-19 Infection.
Brief Title: A Safety and Efficacy Study of Hymecromone Tablets for the Treatment of Patients With COVID-19.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Hao Fang, Chief physician, Vice President, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QJXDS-22-01
Record Dates: First submitted 2022-05-20; First posted 2022-05-23 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
Keywords: COVID-19; Hymecromone
MeSH Terms: conditions — COVID-19 | interventions — Hymecromone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Conventional treatment combined with Hymecromone tablets, 0.4g , tid ac, 7 days.
  Interventions: Drug: Hymecromone tablets
- Control group (Placebo Comparator): Conventional treatment combined with placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Hymecromone tablets — Conventional treatment combined with Hymecromone tablets, 0.4g , tid ac, 7 days.
  Arms: Experimental group
Other: Placebo — Conventional treatment combined with Placebo.
  Arms: Control group

SUMMARY:
The coronavirus (SARS-CoV-2) is a new strain of coronavirus found in human in 2019, which causes epidemic worldwide. A study found that the increase in hyaluronic acid levels is closely related to the clinical symptoms of COVID-19, including pulmonary ground glass lesions, lymphocytopenia, immune response and cytokine storms, systemic vascular diseases, thrombotic coagulation disorders, which suggests that hyaluronic acid could be an important target for COVID-19 treatment and could improve the clinical symptoms of COVID-19 patients.

The results from a recent clinical trial recruited 144 patients with COVID-19 show that the inhibitor of hyaluronic acid synthesis, hymecromone, can significantly improve clinical symptoms, such as lung lesions and lymphocytopenia in COVID-19 patients. Therefore, hymecromone has the potential to become one of the options of COVID-19 treatment.

This study is a single-center, randomized, parallel controlled, double-blind clinical trial designed to evaluate the efficacy and safety of Hymecromone tablets in subjects aged 18-90 years (with boundary values) with a confirmed mild or moderate form of COVID-19 infection. The aim of this study is to optimize the program of the combination of hymecromone in the treatment of COVID-19 to improve the therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have a positive SARS-CoV-2 test result ;
2. Participants who have been diagnosed with mild or ordinary type of COVID-19 infection;
3. Participants whose serum hyaluronic acid level was higher than the upper limit of normal value;
4. Participants who must agree to adhere to contraception restrictions;
5. Participants who understand and agree to comply with planned study procedures;
6. Participants who give signed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Participants who have any of the following conditions when screening:

   1. ALT or AST > 5 ULN;
   2. Scr > 1.5 ULN or Ccr < 50 mL/min;
   3. TBIL > 2ULN ;
   4. HGB ≤ 90 g/ L;
   5. PLT ≤ 75×10^9/ L;
2. Participants who have suspected/active infections during the screening period including uncontrolled active bacterial, viral or fungal infections that require systemic treatment, except COVID-19 virus infections;
3. Participants who have any active autoimmune diseases during the screening period and need to be treated with immunosuppressants, including biological agents;
4. Participants who have a medical history of organ transplantation, or plan for organ transplantation including liver transplantation;
5. Participants who need a loading dose of anti-platelet drugs, such as aspirin (>300 mg/day) and clopidogrel (>300 mg/day);
6. Participants who have a medical history of central nervous system and digestive system bleeding, or a tendency of gastrointestinal bleeding, local active ulcer lesions included, in the last three months;
7. Participants who have biliary obstruction;
8. Female participants who are pregnant or breast-feeding or plan to be pregnant within this study period;
9. Male participants whose wife or partner plan to be pregnant within this study period.
10. Participants who have taken the drugs containing coumarin compounds, such as warfarin, within 3 days before screening;
11. Participants who have other diseases requiring hospitalization and/or in a need of surgical treatment within 7 days before screening, or have suffered from life-threatening diseases within 30 days before screening;
12. Participants who have known allergies to any of the components used in the formulation of the interventions;
13. Participants who have taken a part in a clinical study of an investigational intervention in the last 28 days. After 5 half-lives or 28 days, whichever is longer, can be allowed for screening;
14. Participants who are not suitable for this trial, and with any medical condition will compromise their own safety.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects who developed disease progression. | Within 28 days after initial treatment.
  To compare the proportion of subjects in the experimental group and the control group who developed disease progression within 28 days after initial treatment.

SECONDARY OUTCOMES:
The incidence of adverse events and serious adverse events. | The whole test process.
  To compare the incidence of adverse events and serious adverse events related to the study treatment in the experimental group and the control group.
The time gap of COVID-19 virus clearance. | From the beginning of the research to the negative report of COVID-19 nucleic acid.
  To compare the time of virus clearance by COVID-19 virus tests in the experimental group and the control group.
The clinical recovery time of the COVID-19 virus infection-related symptoms. | From the beginning of the research to the disappearance of clinical symptoms.
  To compare the clinical recovery time of the COVID-19 virus infection-related symptoms in the experimental group with the control group.
The change of the serum hyaluronic acid. | Between baseline and the end of study observation.
  To compare the serum hyaluronic acid level between baseline and the end of study observation of all subjects in the experimental group and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Fang, Principal Investigator — Zhong Shan Hospital affiliated to Fudan University
Locations (1):
- Zhong Shan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang S, Ling Y, Zhao F, Li W, Song Z, Wang L, Li Q, Liu M, Tong Y, Chen L, Ru D, Zhang T, Zhou K, Zhang B, Xu P, Yang Z, Li W, Song Y, Xu J, Zhu T, Shan F, Yu W, Lu H. Hymecromone: a clinical prescription hyaluronan inhibitor for efficiently blocking COVID-19 progression. Signal Transduct Target Ther. 2022 Mar 18;7(1):91. doi: 10.1038/s41392-022-00952-w. PMID 35304437
- [Background] Li W, Yang S, Xu P, Zhang D, Tong Y, Chen L, Jia B, Li A, Lian C, Ru D, Zhang B, Liu M, Chen C, Fu W, Yuan S, Gu C, Wang L, Li W, Liang Y, Yang Z, Ren X, Wang S, Zhang X, Song Y, Xie Y, Lu H, Xu J, Wang H, Yu W. SARS-CoV-2 RNA elements share human sequence identity and upregulate hyaluronan via NamiRNA-enhancer network. EBioMedicine. 2022 Feb;76:103861. doi: 10.1016/j.ebiom.2022.103861. Epub 2022 Feb 3. PMID 35124429
- [Background] Nagy N, Kuipers HF, Frymoyer AR, Ishak HD, Bollyky JB, Wight TN, Bollyky PL. 4-methylumbelliferone treatment and hyaluronan inhibition as a therapeutic strategy in inflammation, autoimmunity, and cancer. Front Immunol. 2015 Mar 23;6:123. doi: 10.3389/fimmu.2015.00123. eCollection 2015. PMID 25852691
- [Derived] Salman L, Martinez L, Faddoul G, Manning C, Ali K, Salman M, Vazquez-Padron R. Hyaluronan Inhibition as a Therapeutic Target for Diabetic Kidney Disease: What Is Next? Kidney360. 2023 Jun 1;4(6):e851-e860. doi: 10.34067/KID.0000000000000126. Epub 2023 Apr 14. PMID 37055910